CLINICAL TRIAL: NCT03812172
Title: Screening for Cardiac Amyloidosis With Nuclear Cardiology for Minority Populations
Brief Title: Screening for Cardiac Amyloidosis With Nuclear Imaging for Minority Populations
Acronym: SCAN-MP
Status: Completed | Type: Observational
Sponsor: Mathew S. Maurer, MD (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Boston Medical Center (Other); Harlem Hospital Center (Other); The Scripps Research Institute (Other); Yale University (Other)
Responsible Party: Sponsor-Investigator, Mathew S. Maurer, MD, Arnold and Arlene Goldstein Professor of Cardiology, Columbia University
Organization: Columbia University (Other)
Other Study IDs: AAAS4054; R01HL139671-01A1 (NIH)
Record Dates: First submitted 2019-01-10; First posted 2019-01-23 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Amyloid Cardiomyopathy, Transthyretin-Related
Keywords: Heart Failure; Cardiac Amyloidosis; TTR mutation; Blacks; Hispanics; Aging
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants in this study provided samples of blood which were analyzed for specific biomarkers and stored for possible future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blacks/Hispanics with Heart Failure: Blacks/Hispanics with heart failure due to transthyretin cardiac amyloidosis were identified by 99mTc-PYP (or 99mTc-HDP) scintigraphy. Those with transthyretin cardiac amyloidosis were further subtyped into those with a genetic cause (ATTRv) and those with a non-genetic cause (ATTRwt - wild type transthyretin cardiac amyloidosis).
  Interventions: Drug: 99mTc-PYP or 99m Tc-HDP

INTERVENTIONS:
Drug: 99mTc-PYP or 99m Tc-HDP — 10-25 mCi of 99mTc-PYP (or 99m Tc-HDP) was administered intravenously and imaging was performed after 3 hours.
  Other Names: Technetium-99m-Pyrophosphate or Technetium-99m-HydroxyMethyleneDiphosphonate

SUMMARY:
In this study, the investigators recruited a cohort of elderly Black and Hispanic patients with heart failure to define the number of patients who have cardiac amyloidosis by utilizing highly sensitive heart imaging and blood tests. The investigators also explored differences in genetics and sex as they relate to heart failure disease progression in cardiac amyloidosis.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) disproportionately afflicts older Black and Hispanic Americans. Transthyretin cardiac amyloidosis (ATTR CA) is caused by myocardial deposition of misfolded transthyretin (TTR or prealbumin) protein and is classified by the genetics of TTR into wild-type (ATTRwt) or hereditary (hATTR or ATTRv). ATTR CA, irrespective of genotype, is an age-dependent, often unrecognized, mechanism underlying HFpEF. While hATTR CA results from point mutations that promote TTR misfolding and amyloid aggregation, factors that contribute to ATTRwt CA are not well defined. While previously thought to be untreatable, promising therapies that have been recently reported are most effective if administered early in disease course. Only a small proportion of individuals with wild-type TTR will develop ATTRwt CA, overwhelmingly reported in Caucasian males beyond age 60 years. However, as an autosomal protein, allele distribution is not sex specific. For hATTR, a substitution of isoleucine for valine (Val142Ile) is the most frequent TTR mutation in the US, observed almost exclusively in Black Americans with an allele frequency of 3.4%. But there are no data regarding the prevalence of ATTRwt CA in African Americans and no data for ATTR CA prevalence, irrespective of genotype, in the Hispanic population. One of the reasons for the knowledge deficit is the challenge of diagnosis. Endomyocardial biopsy, while nearly 100% sensitive and specific, is impractical as a screening test and genotyping alone of patients is insufficient to identify ATTR CA because wild-type patients develop disease. In this study, the investigators used a highly accurate technique for ATTR CA identification using Tc99m-pyrophosphate (PYP) imaging that avoids the need for biopsy. (Tc99m-HDP may have been used in cases of interrupted supply of PYP) Tc99m-PYP myocardial uptake can occur before echocardiographic or clinical changes, suggesting enhanced sensitivity. While studies using the technique have suggested that 10-15% of elderly hospitalized patients with heart failure may have ATTR CA, Tc99m-PYP had not been applied broadly in heart failure patients as a means to facilitate early diagnosis. The overall hypothesis is that a significant proportion of heart failure in elderly Blacks and Hispanics is caused ATTR CA. Using these non-invasive tests, the investigators will establish the prevalence of ATTR CA.

ELIGIBILITY:
Inclusion Criteria:

1. Black or Hispanic of Caribbean origin.
2. Age ≥ 60 years.
3. Diagnosis of heart failure, confirmed by one of two methods:

   1. Modified criteria utilized by Rich et al. which include a history of acute pulmonary edema or the occurrence of at least two of the following that improved with diuretic therapy without another identifiable cause: dyspnea on exertion, paroxysmal nocturnal dyspnea, orthopnea, bilateral lower extremity edema or exertional fatigue, and
   2. National Health and Nutrition Examination Survey (NHANES) congestive heart failure (CHF) criteria with a score ≥3.
4. Left ventricular septal OR inferolateral wall thickness ≥12 mm by echocardiography.
5. Left ventricular Ejection fraction >30% by echocardiography.
6. Able to understand and sign the informed consent document after the nature of the study has been fully explained.

Exclusion Criteria:

1. Primary amyloidosis (AL) or secondary amyloidosis (AA).
2. Prior liver or heart transplantation.
3. Active malignancy or non-amyloid disease with expected survival of less than 1 year.
4. Heart failure, in the opinion of the investigator, primarily caused by severe left-sided valve disease. Note: if valve was repaired, subject may be considered as no longer with severe valve disease.Heart failure, in the opinion of the investigator, primarily caused by either valve disease or ischemic heart disease.
5. Heart failure, in the opinion of the investigator, primarily caused by ischemic heart disease.
6. Ventricular assist device or anticipated within the next 6 months.
7. Impairment from stroke, injury or other medical disorder that precludes participation in the study.
8. Disabling dementia or other mental or behavioral disease.
9. Enrollment in a clinical trial not approved for co-enrollment.
10. Expected use of continuous intravenous inotropic therapy in the next 6 months.
11. High risk for non-adherence as determined by screening evaluation.
12. Inability or unwillingness to comply with the study requirements.
13. Chronic kidney disease with eGFR <15 mL/min/1.73 m2 or ESRD.
14. Weight >350 lb.
15. Nursing home resident.
16. Other reason that would make the subject inappropriate for entry into this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Blacks and Caribbean Hispanics with heart failure not primarily due to ischemic heart disease or valvular disease.
Sampling Method: Probability Sample
Enrollment: 646 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathew S. Maurer, MD, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - Yale University/Yale New Haven Medical Center, New Haven, Connecticut
  - Boston Medical Center/Boston University Medical Center, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York
  - Harlem Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maurer MS, Schwartz JH, Gundapaneni B, Elliott PM, Merlini G, Waddington-Cruz M, Kristen AV, Grogan M, Witteles R, Damy T, Drachman BM, Shah SJ, Hanna M, Judge DP, Barsdorf AI, Huber P, Patterson TA, Riley S, Schumacher J, Stewart M, Sultan MB, Rapezzi C; ATTR-ACT Study Investigators. Tafamidis Treatment for Patients with Transthyretin Amyloid Cardiomyopathy. N Engl J Med. 2018 Sep 13;379(11):1007-1016. doi: 10.1056/NEJMoa1805689. Epub 2018 Aug 27. PMID 30145929
- [Background] Castano A, Haq M, Narotsky DL, Goldsmith J, Weinberg RL, Morgenstern R, Pozniakoff T, Ruberg FL, Miller EJ, Berk JL, Dispenzieri A, Grogan M, Johnson G, Bokhari S, Maurer MS. Multicenter Study of Planar Technetium 99m Pyrophosphate Cardiac Imaging: Predicting Survival for Patients With ATTR Cardiac Amyloidosis. JAMA Cardiol. 2016 Nov 1;1(8):880-889. doi: 10.1001/jamacardio.2016.2839. PMID 27557400
- [Background] Gillmore JD, Maurer MS, Falk RH, Merlini G, Damy T, Dispenzieri A, Wechalekar AD, Berk JL, Quarta CC, Grogan M, Lachmann HJ, Bokhari S, Castano A, Dorbala S, Johnson GB, Glaudemans AW, Rezk T, Fontana M, Palladini G, Milani P, Guidalotti PL, Flatman K, Lane T, Vonberg FW, Whelan CJ, Moon JC, Ruberg FL, Miller EJ, Hutt DF, Hazenberg BP, Rapezzi C, Hawkins PN. Nonbiopsy Diagnosis of Cardiac Transthyretin Amyloidosis. Circulation. 2016 Jun 14;133(24):2404-12. doi: 10.1161/CIRCULATIONAHA.116.021612. Epub 2016 Apr 22. PMID 27143678
- [Background] Ruberg FL, Maurer MS, Judge DP, Zeldenrust S, Skinner M, Kim AY, Falk RH, Cheung KN, Patel AR, Pano A, Packman J, Grogan DR. Prospective evaluation of the morbidity and mortality of wild-type and V122I mutant transthyretin amyloid cardiomyopathy: the Transthyretin Amyloidosis Cardiac Study (TRACS). Am Heart J. 2012 Aug;164(2):222-228.e1. doi: 10.1016/j.ahj.2012.04.015. PMID 22877808
- [Background] Ruberg FL, Grogan M, Hanna M, Kelly JW, Maurer MS. Transthyretin Amyloid Cardiomyopathy: JACC State-of-the-Art Review. J Am Coll Cardiol. 2019 Jun 11;73(22):2872-2891. doi: 10.1016/j.jacc.2019.04.003. PMID 31171094
- [Background] Maurer MS, Bokhari S, Damy T, Dorbala S, Drachman BM, Fontana M, Grogan M, Kristen AV, Lousada I, Nativi-Nicolau J, Cristina Quarta C, Rapezzi C, Ruberg FL, Witteles R, Merlini G. Expert Consensus Recommendations for the Suspicion and Diagnosis of Transthyretin Cardiac Amyloidosis. Circ Heart Fail. 2019 Sep;12(9):e006075. doi: 10.1161/CIRCHEARTFAILURE.119.006075. Epub 2019 Sep 4. PMID 31480867
- [Background] Kittleson MM, Maurer MS, Ambardekar AV, Bullock-Palmer RP, Chang PP, Eisen HJ, Nair AP, Nativi-Nicolau J, Ruberg FL; American Heart Association Heart Failure and Transplantation Committee of the Council on Clinical Cardiology. Cardiac Amyloidosis: Evolving Diagnosis and Management: A Scientific Statement From the American Heart Association. Circulation. 2020 Jul 7;142(1):e7-e22. doi: 10.1161/CIR.0000000000000792. Epub 2020 Jun 1. PMID 32476490
- [Derived] Ruberg FL, Teruya S, Helmke S, Smiley DA, Fine D, Kurian D, Raiszadeh F, Prokaeva T, Spencer B, Wong S, Pandey S, Blaner WS, DeLuca A, Johnson LL, Kinkhabwala MP, Leb J, Mintz A, LaValley MP, Einstein AJ, Cohn E, Gallegos C, Murtagh G, Kelly JW, Miller EJ, Maurer MS. Transthyretin Cardiac Amyloidosis in Older Black and Hispanic Individuals With Heart Failure. JAMA Cardiol. 2025 Oct 1;10(10):1034-1043. doi: 10.1001/jamacardio.2025.2948. PMID 40928765
- [Derived] Madhani A, Sabogal N, Massillon D, Paul LD, Rodriguez C, Fine D, Helmke S, Winburn M, Kurian D, Raiszadeh F, Teruya S, Cohn E, Einstein AJ, Miller EJ, Connors LH, Maurer MS, Ruberg FL. Clinical Penetrance of the Transthyretin V122I Variant in Older Black Patients With Heart Failure: The SCAN-MP (Screening for Cardiac Amyloidosis With Nuclear Imaging in Minority Populations) Study. J Am Heart Assoc. 2023 Aug;12(15):e028973. doi: 10.1161/JAHA.122.028973. Epub 2023 Jul 24. PMID 37486082
- [Derived] Ruberg FL, Blaner WS, Chiuzan C, Connors LH, Einstein AJ, Fine D, Helmke S, Kurian D, Pandey S, Raiszadeh F, Rodriguez C, Sabogal N, Teruya S, Winburn M, Chung WK, Cohn E, Miller EJ, Kelly JW, Maurer MS. Design and Rationale the SCAN-MP (Screening for Cardiac Amyloidosis With Nuclear Imaging in Minority Populations) Study. J Am Heart Assoc. 2023 Apr 18;12(8):e028534. doi: 10.1161/JAHA.122.028534. Epub 2023 Apr 17. PMID 37066788

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Black and Hispanic Caribbean patients with heart failure were recruited from North Manhattan (NYP West and Harlem Hospitals), Boston and New Haven via academic research facilities at Columbia University Irving Medical Center, Boston Medical Center and Yale/New Haven Health Center from 5-19-2019 until 6-12-2024
Groups:
- Self-Identified Black Race Participants With Heart Failure: ATTR-CA prevalence among subjects with heart failure self-identified as Black within predefined categories, (i.e., overall, men, women, Hispanic ethnicity age ≤75 and age >75)
  Transthyretin cardiac amyloidosis status was determined by 99mTc-PYP (or 99mTc-HDP) scintigraphy.
  Those with transthyretin cardiac amyloidosis were further subtyped into those with a genetic cause (ATTRv) variant transthyretin cardiac amyloidosis and those with a non-genetic cause (ATTRwt - wild-type transthyretin cardiac amyloidosis).
- Self-identified Non-Black Participants With Heart Failure:: ATTR-CA prevalence among subjects with heart failure not self-identified as Black within predefined categories, (i.e., overall, men, women, Hispanic ethnicity age ≤75 and age >75)
  Transthyretin cardiac amyloidosis status was determined by 99mTc-PYP (or 99mTc-HDP) scintigraphy.
  Those with transthyretin cardiac amyloidosis were further subtyped into those with a genetic cause (ATTRv) variant transthyretin cardiac amyloidosis and those with a non-genetic cause (ATTRwt - wild-type transthyretin cardiac amyloidosis).
Period: Overall Study
Arm/Group | Self-Identified Black Race Participants With Heart Failure | Self-identified Non-Black Participants With Heart Failure:
Started | 550 | 96
Completed | 550 | 96
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: In follow-up to initial screening visit subjects who were determined to have ATTR-CA or the v142i variant without diagnosis of ATTR-CA (by PYP or HMDP scan) were asked to return for measurement of biomarkers, self-assessment questionnaires and functionality measures at 6 and 12 months, plus echo at 12 months. Subjects who were not found to have either ATTR-CA or v142i variant were followed up only by phone or chart review to determine outcomes.
Groups:
- Self-Identified as Black, Subjects With Heart Failure: ATTR-CA prevalence among subjects with heart failure self-identified as Black within predefined categories, (i.e., overall, men, women, Hispanic ethnicity age ≤75 and age >75)
  Transthyretin cardiac amyloidosis status was determined by 99mTc-PYP (or 99mTc-HDP) scintigraphy.
  Those with transthyretin cardiac amyloidosis were further subtyped into those with a genetic cause (ATTRv - variant transthyretin cardiac amyloidosis) and those with a non-genetic cause (ATTRwt - wild-type transthyretin cardiac amyloidosis).
- Self-identified as Non-Black, Subjects With Heart Failure: ATTR-CA prevalence among subjects with heart failure not self-identified as Black within predefined categories, (i.e., overall, men, women, Hispanic ethnicity age ≤75 and age >75)
  Transthyretin cardiac amyloidosis status was determined by 99mTc-PYP (or 99mTc-HDP) scintigraphy.
  Those with transthyretin cardiac amyloidosis were further subtyped into those with a genetic cause (ATTRv - variant transthyretin cardiac amyloidosis) and those with a non-genetic cause (ATTRwt - wild-type transthyretin cardiac amyloidosis).
- Total: Total of all reporting groups
Arm/Group | Self-Identified as Black, Subjects With Heart Failure | Self-identified as Non-Black, Subjects With Heart Failure | Total
Number analyzed (Participants) | 550 | 96 | 646
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 118 | 16 | 134
  >=65 years | 432 | 80 | 512
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 282 | 45 | 327
  Male | 268 | 51 | 319
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 90 | 96 | 186
  Not Hispanic or Latino | 460 | 0 | 460
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 547 | 0 | 547
  White | 0 | 12 | 12
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 83 | 83

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Transthyretin Cardiac Amyloidosis (ATTR-CA) in Cohort of Caribbean Hispanics and Blacks With Heart Failure (HF)
Description: The prevalence of ATTR cardiac amyloidosis was calculated from among the number of subjects within the cohort determined to be ATTR-CA positive. Determination of ATTR-CA was defined as significant myocardial retention of Tc-99 PYP. The prevalence is expressed as a percentage of total enrollment.
  ATTR-CA prevalence is reported for two different groups: Self-identified as Black, subjects with Heart Failure and Self-identified as non-Black, subjects with Heart Failure.
Time Frame: Study Participation of One Year
Measure: Number; unit: percentage of participants
Groups:
- Self-identified as Black, Subjects With Heart Failure: ATTR-CA prevalence, among subjects with heart failure who self-identified as Black, which was determined by 99mTc-PYP (or 99mTc-HDP) scintigraphy.
- Self-identified as Non-Black, Subjects With Heart Failure: ATTR-CA prevalence, among subjects with heart failure who did not self-identify as Black, which was determined by 99mTc-PYP (or 99mTc-HDP) scintigraphy.
Arm/Group | Self-identified as Black, Subjects With Heart Failure | Self-identified as Non-Black, Subjects With Heart Failure
Number analyzed (Participants) | 550 | 96
percentage of participants | 7.8 | 0

2. Primary Outcome: Age Distribution of ATTR Cardiac Amyloidosis
Description: The prevalence of ATTR cardiac amyloidosis was calculated from among the number of subjects within the cohort determined to be ATTR-CA positive among participants ≤75 years or >75 years enrolled in this study. Determination of ATTR was defined as significant myocardial retention of Tc-99 PYP. The prevalence is expressed as a percentage of total enrollment.
  ATTR-CA prevalence is reported for two different groups: Self-identified as Black, subjects with Heart Failure and Self-identified as non-Black, subjects with Heart Failure.
Time Frame: Study Participation of One Year
Population: Data is separately provided for the study population who were ≤75 years and those who were >75 years old.
Measure: Number; unit: percentage of participants
Groups:
- Self-identified as Black, Subjects With Heart Failure: ATTR-CA prevalence, among subjects with heart failure who self-identified as Black stratified by age group </= 75 years or >75years, which was determined by 99mTc-PYP (or 99mTc-HDP) scintigraphy.
- Self-identified as Non-Black, Subjects With Heart Failure: ATTR-CA prevalence, among subjects with heart failure who did not self-identify as Black (stratified by age group </= 75 years or >75years) due to transthyretin cardiac amyloidosis which was determined by 99mTc-PYP (or 99mTc-HDP) scintigraphy.
Arm/Group | Self-identified as Black, Subjects With Heart Failure | Self-identified as Non-Black, Subjects With Heart Failure
Number analyzed (Participants) | 550 | 96
percentage of participants
  Subjects ≤75 years: number analyzed (Participants) | 322 | 51
  Subjects ≤75 years | 3.42 | 0
  Subjects >75 years: number analyzed (Participants) | 228 | 45
  Subjects >75 years | 14.04 | 0

3. Primary Outcome: Sex Distribution of ATTR Cardiac Amyloidosis
Description: The prevalence of ATTR cardiac amyloidosis was calculated from among the number of subjects within the cohort determined to be ATTR-CA positive among male and female participants enrolled in this study. Determination of ATTR was defined as significant myocardial retention of Tc-99 PYP. The prevalence is expressed as a percentage of total enrollment.
  ATTR-CA prevalence is reported for two different groups: Self-identified as Black, subjects with Heart Failure and Self-identified as non-Black, subjects with Heart Failure.
Time Frame: Study Participation of One Year
Population: Data is separately provided for the study population who were male and those who were female.
Measure: Number; unit: percentage of participants
Arm/Group | Self-identified as Black, Subjects With Heart Failure | Self-identified as Non-Black, Subjects With Heart Failure
Number analyzed (Participants) | 550 | 96
percentage of participants
  Percentage of Male participants with ATTR: number analyzed (Participants) | 268 | 51
  Percentage of Male participants with ATTR | 9.7 | 0
  Percentage of female participants with ATTR: number analyzed (Participants) | 282 | 45
  Percentage of female participants with ATTR | 6 | 0

4. Primary Outcome: Self-Identified Hispanic Ethnicity Distribution of ATTR Cardiac Amyloidosis.
Description: The prevalence of ATTR cardiac amyloidosis was calculated from among the number of subjects within the cohort determined to be ATTR-CA positive among those self-identified as Hispanic, enrolled in this study. Determination of ATTR was defined as significant myocardial retention of Tc-99 PYP. The prevalence is expressed as a percentage of total enrollment.
  ATTR-CA prevalence is reported for two different groups: Self-identified as Black, subjects with Heart Failure and Self-identified as non-Black, subjects with Heart Failure.
Time Frame: Study Participation of One Year
Measure: Number; unit: percentage of participants
Arm/Group | Self-identified as Black, Subjects With Heart Failure | Self-identified as Non-Black, Subjects With Heart Failure
Number analyzed (Participants) | 90 | 96
percentage of participants | 4.4 | 0

5. Primary Outcome: ATTR Type Distribution of Cardiac Amyloidosis
Description: The prevalence of ATTR cardiac amyloidosis was calculated from among the number of subjects within the cohort determined to be ATTR-CA positive among those variant (v142i) and non-variant (wild-type) participants enrolled in this study. Determination of ATTR was defined as significant myocardial retention of Tc-99 PYP. The prevalence is expressed as a percentage of total enrollment.
  ATTR-CA prevalence is reported for two different groups: Self-identified as Black, subjects with Heart Failure and Self-identified as non-Black, subjects with Heart Failure.
Time Frame: Study Participation of One Year
Measure: Count of Participants; unit: Participants
Arm/Group | Self-identified as Black, Subjects With Heart Failure | Self-identified as Non-Black, Subjects With Heart Failure
Number analyzed (Participants) | 550 | 96
Participants
  Subjects with v142i variant | 19 | 0
  Subjects without v142i variant | 24 | 0

ADVERSE EVENTS:
Time Frame: One Year
Description: Only adverse events that met the specified criteria listed in the protocol were collected. The protocol states: "In accordance with 21 CFR 312.32(a), a suspected adverse reaction (SAR) means any adverse event for which there is a reasonable possibility that the drug caused the adverse event." Therefore only events adjudged to be related to PYP administration are listed.
Groups:
- Self Identified as Black, Subjects With Heart Failure: Adverse event prevalence, among subjects with heart failure who self-identified as Black, according to description above.
- Self Identified as Non-Black, Subjects With Heart Failure: Adverse event prevalence, among subjects with heart failure who self-identified as non-Black, according to description above.
Arm/Group | Self Identified as Black, Subjects With Heart Failure | Self Identified as Non-Black, Subjects With Heart Failure
All-Cause Mortality (participants affected / at risk) | 22/550 | 9/96
Serious Adverse Events (participants affected / at risk) | 0/550 | 0/96
Other Adverse Events (participants affected / at risk) | 2/550 | 0/96
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Self Identified as Black, Subjects With Heart Failure (N=550) | Self Identified as Non-Black, Subjects With Heart Failure (N=96)
Nausea (Gastrointestinal disorders) | 1 (1) | 0
Dizziness (General disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT03812172/Prot_SAP_000.pdf